CLINICAL TRIAL: NCT06732557
Title: Muscle Energy Technique Versus Mulligan Mobilization on Forward Head Posture: a Randomized Controlled Trial
Brief Title: Muscle Energy Technique Versus Mulligan Mobilization on Forward Head Posture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Nazih Radwan Meshref, teaching assistant of Basic Science Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005077
Record Dates: First submitted 2024-12-07; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture
Keywords: forward head posture; Mulligan Mobilization; Muscle energy technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Control group (Traditional treament) (Sham Comparator): patients will receive traditional treatment (isometric exercise for deep neck flexors plus sub occipital release).
  Interventions: Other: Traditional treatments
- Group B (muscle energy technique group) (Experimental): Patients will receive muscle energy Technique for upper trapezius, elevator scapulae and sternocleidomastoid
  Interventions: Other: Traditional treatments; Other: muscle energy technique
- Group C (Mulligan Mobilization Group) (Active Comparator): Patients will receive Mulligan mobilization
  Interventions: Other: Traditional treatments; Other: Mulligan Mobilization

INTERVENTIONS:
Other: Traditional treatments — Isometric exercise for deep neck flexors and sub occipital release
Other: muscle energy technique — Muscle energy technique for upper trapezius, elevator scapulae and sternocleidomastoid
  Arms: Group B (muscle energy technique group)
Other: Mulligan Mobilization — Mulligan mobilization in the form of SNAGS for rotation, lateral flexion, extension and flexion
  Arms: Group C (Mulligan Mobilization Group)

SUMMARY:
sixty patients with forward head posture will be randomized to three groups Group A: will receive traditional treatment ( isometric exercise for deep neck flexors plus sub occipital release).

Group B: will receive traditional treatment plus muscle energy technique for upper trapezius, elevator scapulae and sternocleidomastoid.

Group C: will receive traditional treatment plus mulligan mobilization

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 45 years
* Non specific neck pain reproduced by neck movement
* Neck pain at least within the last three months
* Limitation in cervical range of motion

Exclusion Criteria:

* cervical spine surgery or injury
* neurologic deficits, infection or inflammation
* cervicogenic headache

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Pain | Before the first session and at the end of the treatment program ( one month)
  Pain will be measured by visual analogue scale which is a valid and reliable scale for measuring pain starts with zero (represents no pain) and ends with 10 (represents maximum pain).
Cervical range of motion | Before the first session and after the end of the treatment program ( one month)
  Cervical range of motion in will be measured by cervical range of motion basic assessment device (CROM) the angle of cervical range of motion will be recorded in degrees to determine the limitation in range of motion
Disability measurement | Before the first session and after the end of the treatment program ( one month)
  Disability will be measured by neck disability index(NDI) is a valid and reliable scale.
  The NDI consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation.
  Scoring: Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst. Alternately, the score can be reported from 0-100. The score is often reported as a percentage (0-100%).
Cervicovertebral angle | Before the first session and after the end of the treatment program ( one month)
  Cervicovertebral angle (CVA) Will be measure by kinovea:
  Normal range is between 55 and 86, If the angle is less than 50 degrees, it will be considered to be FHP. Adhesive markers (8 mm in diameter) will be placed on the participant's C7 spinous process and tragus of the ear. The physical therapist will observe the participant from the lateral side while standing and then take a picture of the participant from a fixed distance (75 cm) and height (150 cm), then with the help of an application sealed by a password which is called KINOVEA, the angle will be measured by placing each vector as following a line from the tragus of the ear to the C7 spinous process and another horizontal line through the C7 spinous. The angle will be recorded in degrees

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://journals.lww.com/ijpt/fulltext/2021/03020/immediate_effect_of_mulligan_s_mobilization_with.10.aspx